CLINICAL TRIAL: NCT05994131
Title: A Multicenter, Open-label, Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerance, Pharmacokinetics and Anti-tumor Efficacy of IN10018 Combined With Third-generation EGFR-TKI in Patients With Advanced EGFR Mutation-positive NSCLC
Brief Title: IN10018 Combination Therapy in Advanced EGFR Mutation-positive NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-014
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: NSCLC
Keywords: EGFR mutation-positve
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group in cohort 1, cohort 2, and cohort 3 (Experimental): IN10018+Furmonertinib
  Interventions: Drug: IN10018; Drug: Furmonertinib
- Control Group in cohort 3 (Active Comparator): Furmonertinib
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: IN10018 — orally taken once daily
  Other Names: BI 853520
  Arms: Experimental Group in cohort 1, cohort 2, and cohort 3
Drug: Furmonertinib — orally taken once daily

SUMMARY:
This is a multicenter, open-label, phase Ib/II clinical study to evaluate the safety, tolerability, pharmacokinetics and antitumor efficacy of IN10018 in combination with third-generation EGFR-TKI (Furmonertinib is the proposed) in previously-treated or naïve advanced EGFR-mutation positive NSCLC.

DETAILED DESCRIPTION:
This study includes 2 parts: Phase Ib-Dose Confirmation and Phase II-Dose Expansion. And 3 cohorts are set up in this study as cohort 1 to enroll subjects currently accepting third-generation EGFR-TKI (Furmonertinib is proposed) as first-line treatment, cohort 2 to enroll subjects who previously accepted third-generation EGFR-TKI treatment and 1-2 lines chemotherapy, and cohort 3 to enroll treatment-naive advanced EGFR mutation-positive NSCLC subjects.

The phase Ib-dose confirmation part will be conducted in cohort 2 and aim to determine the recommended phase II dose (RP2D) of IN10018 in combination with Furmonertinib. Phase II-Dose Expansion part will be conducted in cohort 1-3 and further explore the antitumor efficacy, safety and PK of IN10018 in combination with Furmonertinib in subjects with previously-treated or naïve advanced EGFR mutation-positive NSCLC.

ELIGIBILITY:
Inclusion Criteria

1. Be able to understand and be willing to sign informed consent.
2. Male or female aged ≥ 18 years old at the time of signing informed consent.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC, who is not suitable for radical surgery or radiotherapy.
4. Documented EGFR mutations known to be associated with EGFR-TKI sensitivity, including Ex19del or L858R. Except for EGFR-TKI sensitive mutation, coexisting with other EGFR mutation types such as T790M can be allowed.
5. Prior systemic antitumor therapy allowed are listed as follows:

   * Cohort 1: Subjects who are on the treatment of Furmonertinib as the first-line treatment setting.
   * Cohort 2: Subjects failed in third-generation EGFR-TKI treatment and also failed in or were intolerant to 1-2 lines of chemotherapy.
   * Cohort 3: subjects who haven't accepted any systemic therapy before. Prior adjuvant or neoadjuvant chemotherapy is permitted if an interval from the lost dose of adjuvant or neoadjuvant chemotherapy to the first documented PD is >6 months.
6. Measurable lesions at baseline according to RECIST 1.1 criteria.
7. Has an ECOG performance status of 0 or 1.
8. Estimated life expectancy is more than 3 months.
9. Adequate bone marrow, liver, renal, and coagulation function within 7 days prior to the first dose of study treatment/randomization.

Exclusion Criteria

1. Have experienced major surgical procedures or major trauma within 28 days prior to the first dose of study treatment/randomization.
2. Have received the following prior systemic antitumor therapy:

   * Cohort 1: Have received chemotherapy, target therapy besides Furmonertinib, immunotherapy, biological therapy, and other antitumor drugs.
   * Cohort 2: Have received chemotherapy, targeted therapy, immunotherapy, biological therapy, and other antitumor drugs within 28 days prior to the first dose of study treatment.
   * Cohort 3: Have received systemic antitumor therapy for locally-advanced or metastatic NSCLC including chemotherapy, target therapy, immunotherapy, biotherapy, etc.
3. Cohort 2 only： Presence of other gene mutations, including ALK mutation, MET amplification, HER2 amplification, RAS mutation, etc. after progression on prior third-generation EGFR-TKI treatment.
4. Cohort 3 only：Has received the treatment of EGFR-TKI。
5. Prior FAK inhibitors treatment.
6. Have received systemic administration of potent inhibitors/inducers of CYP3A4, or P-gp inhibitors within 14 days prior to the first dose of treatment/randomization or are expected to receive systemic administration of these drugs during study treatment.
7. Has received radiotherapy for study disease or radiotherapeutic area covered for more than 30% of the bone marrow within 28 days prior to the first dose of study treatment/randomization.
8. Has had interstitial lung disease (ILD), drug-induced ILD, radiation pneumonia requiring steroid therapy; or diagnosis of clinically active ILD during the screening period.
9. Has a prior history of other malignancy within 3 years prior to signing informed consent.
10. Has known symptoms of spinal cord compression, active central nervous system (CNS) metastases, and/or carcinomatous meningitis.
11. Has a history of severe cardiovascular or cerebrovascular diseases within 6 months prior to the first dose of study treatment/randomization.
12. Has known uncontrollable pleural effusion, pericardial effusion, and ascites.
13. Has hemoptysis within 1 month prior to the first dose of study treatment/randomization with a blood volume of ≥2.5 mL every time or expected to require continuous hemostasis therapy during the study treatment.
14. Has active infections that are poorly controlled by systemic treatment.
15. Has active tuberculosis.
16. Known allergy, hypersensitivity or intolerance to IN10018 and/or third-generation EGFR-TKI, or their ingredients.
17. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of IN10018 in combination with third-generation EGFR-TKI in subjects with advanced EGFR mutation-positive NSCLC. | 3 years
  Evaluate the number of patients with dose-limited toxicities (DLTs); Determine the RP2D of IN10018 in combination with third-generation EGFR-TKI in subjects with advanced NSCLC.
ORR of IN10018 in combination with third-generation EGFR-TKI in subjects with advanced EGFR mutation-positive NSCLC. | 3 years
  Defined as the proportion of subjects with complete response (CR) or partial response (PR)
Tumor Shrinkage Rate (TSR) of IN10018 in combination with third-generation EGFR-TKI in cohort 3 of advanced treatment-naive EGFR mutation-positive NSCLC. | 3 years
  Defined as the percentage of subjects with the best shrinkage rate of target lesions ≥ 70% and simultaneously with a best response of partial response (PR) or complete response (CR).

SECONDARY OUTCOMES:
PFS of IN10018 in combination with third-generation EGFR-TKI in advanced EGFR mutation-positive NSCLC. | 3 years
  Defined as the time from the first dose of study treatment/randomization to first documentation of disease progression or to death due to any cause, whichever comes first.
DOR of IN10018 in combination with third-generation EGFR-TKI in advanced EGFR mutation-positive NSCLC. | 3 years
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
DCR of IN10018 in combination with third-generation EGFR-TKI in advanced EGFR mutation-positive NSCLC. | 3 years
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
OS of IN10018 in combination with third-generation EGFR-TKI in advanced EGFR mutation-positive NSCLC. | 3 years
  Defined as the time from the first dose of study treatment/randomization to the date of death due to any cause.
Number of patients with adverse event | 3 years
  The number of participants who experienced AEs is presented.
PK: AUC of IN10018 following single dose administration and at steady state | 3 years
  Area under the concentration-time curve (AUC)
PK: Cmax of IN10018 following single dose administration and at steady state | 3 years
  Maximum concentration (Cmax)
PK:Ctrough of IN10018 following single dose administration and at steady state | 3 years
  Trough concentration (Ctrough)
PK:Tmax of IN10018 following single dose administration and at steady state | 3 years
  Time to Cmax (Tmax)
PK:t1/2 of IN10018 following single dose administration and at steady state | 3 years
  Elimination half-life (t1/2).
PK:CL/F of IN10018 following single dose administration and at steady state | 3 years
  apparent clearance (CL/F)
PK:Vd/F of IN10018 following single dose administration and at steady state | 3 years
  Apparent volume of distribution (Vd/F)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No